## **VERBAL INFORMED CONSENT:**

**Study Title:** Comparison of Distally Based Sural Artery and Supramalleolar Flap for Coverage of Dorsum of Foot and Ankle Defects; A CROSS-SECTIONAL STUDY OF 53 PATIENTS

**ERC Ref No:** 4452

**Principal Investigator**: Dr Pervaiz Hashmi, Department of surgery, Aga Khan University Hospital

Other Investigators: Abeer Musaddiq, Dr Muhammad Ali, Dr Zohaib Nawaz

We (investigators) are from the Aga Khan University hospital and calling regarding a study which is being conducted by our hospital. We are conducting this study to analyze the long-term clinical and functional outcomes of lower extremity/extremities after Flap surgery.

You have been invited to participate in this study. You will be asked the specific data via telephone about your Activity of Daily living after Flap Surgery. The survey will take approximately 15-20 minutes of your time. Your identity and any provided information will be kept strictly confidential. However, the study may be published in journal and elsewhere without disclosing your identity. You are free to choose whether to participate or not in this study.

This study has been approved by The Aga Khan University Ethics Review Committee and will be conducted in accordance with the ethical principles.

## **Authorization:**

I have listened and understand the form and I agree to participate in this study.

| Name of Patient/participant: | |
|---------------------------------------------------|---|
| Name and designation of Person obtaining Consent: | |
| Signature of Person obtaining Consent: | |
| Name and designation of Witness: | _ |
| Signature of Witness: | |
| Date: | |